CLINICAL TRIAL: NCT05558826
Title: Analysis of Intra-abdominal Pressure and Trendelenburg Position Effect on Dynamic Indices of Arterial Pressure Waveform
Brief Title: Pressure Analysis of Trendelenburg Position Effect on Indices From Arterial Pressure
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2022-04-002AC
Record Dates: First submitted 2022-09-25; First posted 2022-09-28 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Anesthesia; Fluid and Electrolyte Imbalance; Hemodynamic Instability
Keywords: Goal directed fluid therapy; Arterial waveform analysis; Pneumoperitoneum; Trendelenburg position
MeSH Terms: conditions — Pneumoperitoneum

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: HemoSphere advanced monitoring platform with Acumen Hypotension Prediction Index Software — After induction of anesthesia, intra-arterial catheterization will be done for invasive blood pressure monitoring and blood sampling as routine clinical practice for major laparoscopic surgery. Arterial line will be connected to HemoSphere advanced monitoring platform with Acumen Hypotension Prediction Index Software for arterial pressure waveform analysis. Dynamic indices including pulse pressure variation (PPV), stroke volume variation (SVV), Hypotension Prediction Index (HPI), Dynamic arterial elastance (Eadyn) and dP/dt will be continuously recorded. Changes in levels of intra-abdominal pressure and angles of Trendelenburg position will be recorded. Data analysis and statistics will be particularly performed to explore the effects of levels of intra-abdominal pressure and angles of Trendelenburg position on dynamic indices of arterial pressure waveform.

SUMMARY:
Intraoperative fluid management is key component of care for patients undergoing surgery. Hypovolemia and hypervolemia both associate with increased morbidity, length of stay in the intensive care unit and mortality. Thus, maintaining adequate intravascular volume yet avoiding fluid overload is crucial to achieve optimal outcomes. Goal-directed fluid therapy based on arterial pressure waveform analysis is widely used for intraoperative fluid management and have been shown to improve surgical outcomes compared with conventional clinical assessment in several studies. However, dynamic indices of arterial pressure waveform analysis such as pulse pressure variation (PPV) and stroke volume variation (SVV) are altered by certain situations including elevated intra-abdominal pressure and Trendelenburg position. Intravascular fluid status might thus be misinterpreted. Carbon dioxide pneumoperitoneum with increased intra-abdominal pressure and Trendelenburg position are commonly seen in laparoscopic surgeries including colorectal, gynecological, and genitourinary procedures. Understanding how dynamic indices change in these clinical situations are essential for achieving appropriate intraoperative fluid management. This study focus on identifying the effects of different levels of intra-abdominal pressure and angles of Trendelenburg position on dynamic indices of arterial pressure waveform.

DETAILED DESCRIPTION:
In this prospective observational study, the investigators will enroll 100 patients undergoing laparoscopic surgery for medical reason. Anesthetic management and surgery will be performed as usual clinical practice.

The investigators will record the digital data exported from standard monitoring instruments, including electrocardiography, photo-plethysmography , blood pressure, neurological system information (Bispectral index and Density spectral array ), the respiratory gas monitoring (gas analyzer and respiratory waveform) and dynamic indices of arterial pressure waveform analysis (cardiac index, stroke volume variation, pulse pressure variation, hypotension prediction index... etc.) from HemoSphere advanced monitoring platform with Acumen Hypotension Prediction Index Software (Edwards Lifesciences) every 20 seconds.

After anesthesia induction as routine clinical practice, slow IV fluid infusion will be maintained. The patient will be placed in Trendelnburg position with different angles ranging from 0-25 degree. CO2 pneumoperitoneum will be created by surgeons for laparoscopic surgery. Changes in levels of intra-abdominal pressure and angles of Trendelenburg position will be recorded. The recording is ended after emergence when surgery ends. All physiological data and demographic data will be stored in digital media after being de-linked from personal identification.

Data analysis and Statistics will be particularly performed to explore the effects of levels of intra-abdominal pressure and angles of Trendelenburg position on dynamic indices of arterial pressure waveform. Methods including signal processing, modeling, classification will be used.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 20 and 80
* Scheduled for laparoscopic surgery
* American Society of Anesthesiologists (ASA) physical status I to III.

Exclusion Criteria:

* Neurologic or behavioral disorders
* American Society of Anesthesiologists (ASA) physical status ≥ IV
* History of arrhythmia
* Drug abuse or alcoholism
* Resting room air SpO2 < 90%.

Ages: 20 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The investigators plan to enroll patients who will laparoscopic surgery under general anesthesia. These patients will be screened for eligibility.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2023-10-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Stroke volume variation (SVV) | Dynamic indices recorded starting after anesthesia induction, and stopped after emergence when surgery ends
  SVV is the ratio of the maximum (SVmax) SV minus the minimum SV (SVmin) to the mean SV (SVmean), averaged over several respiratory cycles. SVV is an indicator of a patient's position on the Frank-Starling Curve. Studies suggested SVV >10 % is associated with fluid responsiveness. SVV will be obtained and recorded from HemoSphere advanced monitoring platform with Acumen Hypotension Prediction Index Software (Edwards Lifesciences).
Pulse pressure variation (PPV) | Dynamic indices recorded starting after anesthesia induction, and stopped after emergence when surgery ends
  PPV is the ratio of the maximum pulse pressure (systolic blood pressure minus diastolic blood pressure; PPmax) minus the minimum pulse pressure (PPmin) to the mean pulse pressure (PPmean), averaged over several respiratory cycles. PPV is an indicator of a patient's position on the Frank-Starling Curve. Studies suggested PPV >13-15 %is associated with fluid responsiveness. PPV will be obtained and recorded from HemoSphere advanced monitoring platform with Acumen Hypotension Prediction Index Software (Edwards Lifesciences).
Hypotension Prediction Index (HPI) | Dynamic indices recorded starting after anesthesia induction, and stopped after emergence when surgery ends
  The Hypotension Prediction Index (HPI) is a prediction model based on features of arterial pressure waveform. It represents as unitless number from 1 to 100. Greater number suggested higher risk of a hypotension event occurring in the future. HPI will be obtained and recorded from HemoSphere advanced monitoring platform with Acumen Hypotension Prediction Index Software (Edwards Lifesciences).
Dynamic arterial elastance (Eadyn) | Dynamic indices recorded starting after anesthesia induction, and stopped after emergence when surgery ends
  Dynamic arterial elastance (Eadyn) is the ratio of pulse pressure variations (PPV) to stroke volume variations (SVV). Studies have shown Eadyn as a predictor of blood pressure response to fluid resuscitation in hypotension, fluid-responsive patients. Eadyn will be obtained and recorded from HemoSphere advanced monitoring platform with Acumen Hypotension Prediction Index Software (Edwards Lifesciences).
dP/dt | Dynamic indices recorded starting after anesthesia induction, and stopped after emergence when surgery ends
  dP/dT (mmHg/second)is the change of left ventricular pressure over time during isovolemic contraction. It is usually used as a predictor of myocardial contractility.

SECONDARY OUTCOMES:
Bispectral index (BIS) value | BIS monitor are recorded starting from anesthesia induction, and stopped after emergence when surgery ends
  Our study records these parameters on an observational basis. Anesthetic management remains identical regardless of patient participation or not. The recorded BIS value reading is uniform and contains only a unitless number ranging from 0 to 100. Different procedures do not give different units. Spectral analysis of the alpha, beta, gamma, theta and delta features of EEG will be performed. Individual band powers are summed separately.

CONTACTS AND LOCATIONS:
Overall Officials: Chien-Kun Ting, MD.PhD, Study Chair — Department of Anesthesiology, Taipei Veterans General Hospital, Taiwan
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jessen MK, Vallentin MF, Holmberg MJ, Bolther M, Hansen FB, Holst JM, Magnussen A, Hansen NS, Johannsen CM, Enevoldsen J, Jensen TH, Roessler LL, Lind PC, Klitholm MP, Eggertsen MA, Caap P, Boye C, Dabrowski KM, Vormfenne L, Hoybye M, Henriksen J, Karlsson CM, Balleby IR, Rasmussen MS, Paelestik K, Granfeldt A, Andersen LW. Goal-directed haemodynamic therapy during general anaesthesia for noncardiac surgery: a systematic review and meta-analysis. Br J Anaesth. 2022 Mar;128(3):416-433. doi: 10.1016/j.bja.2021.10.046. Epub 2021 Dec 13. PMID 34916049
- [Background] Maheshwari K, Shimada T, Yang D, Khanna S, Cywinski JB, Irefin SA, Ayad S, Turan A, Ruetzler K, Qiu Y, Saha P, Mascha EJ, Sessler DI. Hypotension Prediction Index for Prevention of Hypotension during Moderate- to High-risk Noncardiac Surgery. Anesthesiology. 2020 Dec 1;133(6):1214-1222. doi: 10.1097/ALN.0000000000003557. PMID 32960954
- [Background] Min JH, Lee SE, Lee HS, Chae YK, Lee YK, Kang Y, Je UJ. The correlation between the Trendelenburg position and the stroke volume variation. Korean J Anesthesiol. 2014 Dec;67(6):378-83. doi: 10.4097/kjae.2014.67.6.378. Epub 2014 Dec 29. PMID 25558337
- [Background] Davies SJ, Vistisen ST, Jian Z, Hatib F, Scheeren TWL. Ability of an Arterial Waveform Analysis-Derived Hypotension Prediction Index to Predict Future Hypotensive Events in Surgical Patients. Anesth Analg. 2020 Feb;130(2):352-359. doi: 10.1213/ANE.0000000000004121. PMID 30896602
- [Background] Tavernier B, Robin E. Assessment of fluid responsiveness during increased intra-abdominal pressure: keep the indices, but change the thresholds. Crit Care. 2011;15(2):134. doi: 10.1186/cc10074. Epub 2011 Mar 18. PMID 21457517